CLINICAL TRIAL: NCT04714554
Title: A Two-Part, Open-Label, Fixed-Sequence, Two-Period Crossover Study to Assess the Effects of Erythromycin on the Pharmacokinetics of Relugolix, Estradiol, and Norethindrone After Administration of the Relugolix/Estradiol/Norethindrone Acetate Fixed-Dose Combination Tablet in Healthy Postmenopausal Women and on the Pharmacokinetics of Relugolix After Administration of a Single 120-mg Dose in Healthy Adult Men
Brief Title: A Study of the Effects of Erythromycin on the Pharmacokinetics of Relugolix, Estradiol, and Norethindrone in Healthy Postmenopausal Women and on the Pharmacokinetics of Relugolix in Healthy Adult Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-054
Record Dates: First submitted 2021-01-08; First posted 2021-01-19 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Relugolix; Estradiol; Norethindrone acetate; Erythromycin; Pharmacokinetics; Norethindrone
MeSH Terms: interventions — relugolix; Erythromycin

STUDY DESIGN:
Intervention Model Description: In each study part (Part 1 and Part 2), study treatments will be administered in a fixed (single) sequence, crossover manner in two sequential treatment periods (Treatment Period 1 and Treatment Period 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Relugolix/E2/NETA Plus Erythromycin (Experimental): Treatment Period 1: Healthy premenopausal women will receive a relugolix/E2/NETA (40 mg/1 mg/0.5 mg) alone on Day 1.
  Treatment Period 2: Healthy premenopausal women will receive erythromycin on Day 1 through 12 (500 mg, QID), with co-administration of a single dose of relugolix/E2/NETA (40 mg/1 mg/0.5 mg) with the morning dose of erythromycin on Day 8.
  Interventions: Drug: Relugolix/E2/NETA FDC; Drug: Erythromycin
- Part 2: Relugolix Plus Erythromycin (Experimental): Treatment Period 1: Male participants will receive a single 120-mg dose of relugolix alone on Day 1.
  Treatment Period 2: Male participants will receive erythromycin on Days 1 through 12 (500 mg, QID), with co-administration of a single 120-mg dose of relugolix with the morning dose of erythromycin on Day 8.
  Interventions: Drug: Relugolix; Drug: Erythromycin

INTERVENTIONS:
Drug: Relugolix/E2/NETA FDC — Relugolix/E2/NETA (40 mg/1 mg/0.5 mg) FDC tablet; oral administration.
  Other Names: Rel-CT
  Arms: Part 1: Relugolix/E2/NETA Plus Erythromycin
Drug: Relugolix — Relugolix 120-mg tablets; oral administration.
  Other Names: MVT-601; TAK-385
  Arms: Part 2: Relugolix Plus Erythromycin
Drug: Erythromycin — Erythromycin 500-mg tablets; oral administration.

SUMMARY:
This is a two-part, open-label, fixed-sequence, two-period crossover drug interaction study to assess the potential effects of erythromycin on the pharmacokinetics of relugolix, estradiol (E2), and norethindrone (NET) in healthy postmenopausal women (Part 1) and the pharmacokinetics of relugolix in healthy adult men (Part 2).

DETAILED DESCRIPTION:
Each study part consists of two sequential treatment periods (Treatment Period 1 and Treatment Period 2) in which study participants will receive study treatments in a fixed (single)-sequence, crossover manner. In Part 1 of the study, a single relugolix/E2/norethindrone acetate (NETA) (40 milligrams [mg]/1 mg/0.5 mg) fixed-dose combination (FDC) tablet will be administered alone on Day 1 of Treatment Period 1; in Treatment Period 2, erythromycin will be administered on Day 1 to Day 12 (500 mg, four times daily [QID]) with co-administration of a single FDC tablet with the morning dose of erythromycin on Day 8. In Part 2 of the study, a single 120-mg dose of relugolix will be administered alone on Day 1 of Treatment Period 1; in Treatment Period 2, erythromycin will be administered on Day 1 to Day 12 (500 mg QID) with co-administration of a single 120-mg dose of relugolix with the morning dose of erythromycin on Day 8. There will be a nine-day washout interval between administration of study drug (the FDC tablet [Part 1] or relugolix 120 mg [Part 2]) on Day 1 of Treatment Period 1 and Treatment Period 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Study participant is considered to be medically healthy, based on a clinical evaluation including medical history, physical examinations, clinical laboratory tests, vital sign measurements, and a 12-lead electrocardiogram performed at the screening visit. Specifically, study participants should meet the following requirements at the screening visit:
* Heart/pulse rate of 50 to 90 beats per minute, inclusive;
* Systolic blood pressure of 90 to 139 millimeters of mercury (mmHg) and a diastolic blood pressure of 60 to 89 mmHg, inclusive;
* A QT interval with Fridericia's correction (QTcF, QTcF = QT/RR(0.33)) ≤ 470 milliseconds;
* Normal renal function at the screening visit, defined as an estimated creatinine clearance ≥ 90 milliliters (mL)/minute by the Cockcroft-Gault equation;
* An alanine aminotransferase, aspartate aminotransferase or bilirubin value within normal limits.
* Part 1 only: Study participant is a female between 40 and 65 years of age, inclusive, at the screening visit.
* Part 2 only: Study participant is a male between 18 and 65 years of age, inclusive, at the screening visit.
* Study participant has a body mass index from ≥ 18.5 to ≤ 32.0 (Part 1) or from ≥ 18.5 to ≤ 30.0 (Part 2) (kilograms/square meter), at the screening visit.
* Part 1 only: Study participant is a postmenopausal female defined as 12 months of spontaneous amenorrhea without an alternative medical cause or six weeks status post bilateral oophorectomy (with or without hysterectomy). A serum follicle-stimulating hormone (FSH) ≥ 40 milli-international units/mL is required to confirm postmenopausal status. Note: women who are amenorrheic due to a surgical procedure (hysterectomy without oophorectomy) and are considered physiologically postmenopausal based on FSH values may participate.

Key Exclusion Criteria:

* Study participant has a clinically significant medical or psychiatric condition or disease (acute or chronic) that, as judged by the investigator, would make the study participant ineligible for participation in the study (for example, compromise the study data, limit the study participant's ability to complete and/or participate in the study).
* Study participant has a current condition or history of significant endocrine, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, urologic, immunologic, or neurologic disorders that, as judged by the investigator, would make the study participant ineligible for participation in the study.
* Study participants with a pre-existing condition interfering with normal gastrointestinal anatomy (with the exception of an uncomplicated appendectomy) or motility, hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* Study participant has unconjugated bilirubin values consistent with Gilbert's syndrome or a history of or current gall bladder or bile-duct disease.
* Part 1 only: Study participant has any contraindications to treatment with E2 and NETA, based on medical history:
* Undiagnosed abnormal genital bleeding;
* Known or suspected history of breast cancer;
* Known or suspected estrogen-dependent neoplasia;
* Active deep vein thrombosis, pulmonary embolism, or history of these conditions;
* Active arterial thromboembolic disease (for example, stroke and myocardial infarction), or a history of these conditions;
* Known anaphylactic reaction or angioedema or hypersensitivity to estradiol or norethindrone acetate;
* Known hepatic impairment or disease;
* Known protein C, protein S, or antithrombin deficiency, or other known thrombophilic disorders.
* Study participant has used prescription or non-prescription drugs, including vitamins and dietary or herbal supplements within 14 days (or 5 half-lives, whichever is longer) prior to study drug administration on Day 1 of Treatment Period 1, unless in the opinion of the Sponsor the medication will not interfere with interpretation of study data or compromise the safety of study participants.
* Study participant has used any medication known to be a strong cytochrome P450 3A inducer and/or P glycoprotein inducer within the timeframe prior to study drug administration on Day 1 of Treatment Period 1.
* Part 1 only: Study participant has used medications containing hormonal products, including injectables, within the timeframe prior to study drug administration on Day 1 of Treatment Period 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Area Under The Concentration-time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Of Relugolix Or Other Analytes | Day 8 predose and up to 120 hours postdose at multiple time points during Treatment Period 2 (Study Days 10 to 22)
Maximum Plasma Concentration (Cmax) Of Relugolix Or Other Analytes | Day 8 predose and up to 120 hours postdose at multiple time points during Treatment Period 2 (Study Days 10 to 22)

SECONDARY OUTCOMES:
Overall Incidence Of Adverse Events | 10 Weeks
Predose Trough Plasma Concentrations (Ctrough) Of Erythromycin | Predose on Day 7 and 8 of Treatment Period 2 (Study Days 10 to 22)

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Monitor, Study Director — Myovant Sciences
Locations (1):
- Clinical Pharmacology of Miami, An Evolution Research Group Portfolio Company, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: No